CLINICAL TRIAL: NCT02150382
Title: Effectiveness of a Standardized Protocol-based Treatment Program on Hypertension Control in Rural China.
Brief Title: China Rural Hypertension Control Project 2014
Status: Withdrawn | Type: Observational
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Yingxian Sun, Chief of Department of Cardiology in First Hospital of China Medical University, First Hospital of China Medical University
Other Study IDs: China Medical University
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2014-05

CONDITIONS: Hypertension
Keywords: hypertension; rural; China; protocol-based treatment
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
China Rural Hypertension Control (CRHC) Project is a cluster randomized trial aims to test the effectiveness of a standardized protocol-based treatment program on hypertension control in rural China.

ELIGIBILITY:
Inclusion Criteria:

* Man and women aged 40 years or older.
* Mean systolic blood pressure ≥140 mm Hg and/or diastolic blood pressure ≥90 mm Hg; and/or use of antihypertensive medications.Mean blood pressure is based on three measurements at two separate days at least two days apart and within one month.
* Permanent residents in the study villages.
* Do not plan to emigrate in the next 2 years.

Exclusion Criteria:

* Unable to provide consent.
* Treated for malignant tumor and life expectancy<2 years judged by study physician.
* Pregnancy, currently trying to become pregnant, or of child-bearing potential and not using birth control.
* Diagnosted psychiatric patients.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All study patients will be recruited from rural areas in Liaoyang County from blood pressure screening. Liaoyang County, Liaoning Province is located in Northeast China.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2016-07 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
a composite outcome of cardiovascular disease and all-cause mortality | up to 2-year

SECONDARY OUTCOMES:
Major cardiovascular diseases | up to 2-year
Fatal and non-fatal stroke | up to 2-year
Fatal and non-fatal myocardial infarction | up to 2-year
Hospitalized or treated heart failure | up to 2-year
Cardiovascular death | up to 2-year
Change in mean systolic and diastolic blood pressure | up to 2-year
Proportion of hypertension control | up to 2-year

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of China Medical University, Shenyang, Liaoning, China